CLINICAL TRIAL: NCT02345538
Title: Use of a Perineometer to Assess Resting Pelvic Muscle Tone in Patients With Pelvic Pain
Brief Title: Use of a Perineometer to Assess Pelvic Muscle Tone
Status: Withdrawn | Type: Observational
Why Stopped: Investigator did not start the project in time; study team decided it was not feasible to begin study as resident was soon graduating. No patients enrolled.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00053004
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with Chronic Pelvic Pain: Use of perineometer to measure pelvic resting tone and contraction in women with chronic pelvic pain and determine if resting tone correlates with severity of pain.
- Women without Chronic Pelvic Pain: Use of perineometer to measure pelvic resting tone and contraction in women without chronic pelvic pain

SUMMARY:
The purpose of this study is to establish the range of pelvic floor pressure in groups of women, including women with and without pelvic pain, and compare the change in perineometer measurements between rest and maximum pelvic floor contraction in women with and without pelvic pain. Purpose is also to determine whether resting pelvic floor perineometer measurements correlate with the severity of pain symptoms in women with chronic pelvic pain.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is defined as non-cyclic pelvic pain lasting at least 6 months. Approximately 3-15% of women are affected by CPP. Care of patients with CPP contributes to considerable healthcare costs, accounting for 880 million dollars annually in outpatient visits alone. Although CPP may be multifactorial, many women have a contribution from increased pelvic floor tone. CPP due to increased pelvic floor tone is usually referred to as levator spasm or high tone pelvic floor dysfunction. Levator tenderness and increased pelvic tone may be identified on physical exam. However, physical exam is somewhat subjective and may vary based on the clinician performing the exam. There are currently no validated, objective measures to judge resting pelvic tone, which 1) limits objective assessment in research studies and 2) limits our ability to assess response to new treatment modalities.

The ability to contract the pelvic floor may be assessed during pelvic exam with a Brink's score. However, there are still elements of subjectivity in components of this score and researchers continue to look for an objective measure of pelvic floor muscle tone. The Peritron perineometer device has been shown to correlate well with pelvic floor contraction, based on Brinks scores.Measurements taken with the Peritron device have better inter-rater reliability than other measures of pelvic floor contraction, which makes it an attractive tool for clinical research. However, its use in clinical research is hampered by the lack of normative data with perineometer measurements. Though there are some studies that use the perineometer to assess resting (i.e. non-contracted) pelvic tone after therapies for pelvic pain, there are no studies that assess the typical perineometer measurements in women with levator spasm, and there are no data to guide how these measurements may compare with women having a normal pelvic floor examination. We hypothesize that: 1) Women with high resting pelvic tone perceived on exam will have high perineometer measurements and women with normal pelvic tone on exam will have low perineometer measurements, regardless of whether or not they report pelvic pain. 2) Women with high resting perineometer measurements will have minimal change in perineometer scores between resting and maximum pelvic floor contraction (squeeze). 3) In women with clinical evidence of levator spasm, resting perineometer measurements will correlate with severity of pelvic pain symptoms. We plan to investigate these hypotheses by executing the following specific aims:

Specific Aim 1: To compare clinical assessment of resting pelvic tone with perineometer measurements in a range of women, including those with and without pelvic pain.

Specific Aim 2: To compare the change in perineometer measurements between rest and maximum pelvic floor contraction in women with and without pelvic pain.

Specific Aim 3: To determine whether resting pelvic floor perineometer measurements correlate with the severity of pain symptoms, as measured by short form McGill questionnaire scores and visual analog scale (VAS), in a subset of women with pelvic pain and clinical evidence of levator spasm.

ELIGIBILITY:
Inclusion Criteria:

* being seen in the Duke Urogynecology or Minimally Invasive Gynecology Clinics

Exclusion Criteria:

* botulinum toxin A injection into bladder or pelvic floor musculature within the prior 9 months
* history of GYN or GU malignancy
* chronic use of muscle relaxants
* exam findings that would preclude the ability of the woman to retain the Peritron device (e.g. narrowed introitus or stage III/IV prolapse).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of adult women, seen in an outpatient urogynecology or minimally invasive gynecology clinic, including women with and without pelvic pain.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
measurement of pelvic pressure in the two groups | 1 day
  using the peritron device at rest and maximum squeeze

SECONDARY OUTCOMES:
Brinks score | 1 day
  measurement of maximum kegel strength on clinical exam
Pelvic pain score | 1 day
  quantification of pelvic pain based on visual analog score and short form McGill pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nazema Siddiqui, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No
study withdrawn